CLINICAL TRIAL: NCT03012425
Title: Pilot Study of Cognitive Behavioral Therapy for Insomnia (CBT-I) and Acupuncture for Insomnia and Related Distress Among Cancer Caregivers
Brief Title: Study of Cognitive Behavioral Therapy for Insomnia (CBT-I) and Acupuncture for Insomnia and Related Distress Among Cancer Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hunter College of City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-001
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Insomnia; Related Distress Among Cancer Caregivers
Keywords: Cognitive Behavioral Therapy; Acupuncture; 17-001
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Acupuncture Therapy; Surveys and Questionnaires

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (CBT-I) (Experimental): Session 1- Review of initial sleep diary, formulation of impression of type/subtype of insomnia, determine modifiable factors, address immediate concerns about participation, discuss motivation & compliance. Session 2- Review of sleep diary, present 4-P model of insomnia, prescribe Sleep Restriction & Stimulus Control Therapy. Session 3- Review of sleep diary, continue with stimulus control & sleep restriction procedures, review of sleep hygiene. Session 4- Review of sleep diary, continue with stimulus control & sleep restriction procedures, introduce & practice relaxation strategies. Session 5- Review of sleep diary, continue with stimulus control & sleep restriction procedures, conduct cognitive therapy to address dysfunctional thoughts underlying insomnia. Session 6- Review of sleep diary, continue with stimulus control & sleep restriction procedures Session 7- Review of sleep diary & overall progress, discuss relapse prevention, further sleep restriction guidelines & prophylaxis.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I); Behavioral: questionnaires; Other: Diurnal Cortisol
- Acupuncture (Experimental): Session 1 - Detailed history and examination, introduction to acupuncture. Sessions 2 - 10 - Each session will begin with insertion and manipulation of needles, which will remain in place for 30 minutes.
  Interventions: Procedure: Acupuncture; Behavioral: questionnaires; Other: Diurnal Cortisol

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
  Arms: Cognitive Behavioral Therapy for Insomnia (CBT-I)
Procedure: Acupuncture
  Arms: Acupuncture
Behavioral: questionnaires
Other: Diurnal Cortisol — saliva test

SUMMARY:
The other aim of this study is to determine which of those two treatments (acupuncture or cognitive behavioral therapy) works better for treating insomnia in Informal Caregivers of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* As per self report, age 18 and older
* As per self report, identifying as an informal caregiver to MSKCC patients of any site or stage of cancer
* Score greater than 7 on the Insomnia Severity Index and meet the criteria for Insomnia Disorder as defined by the Diagnostic and Statistical Manual of Mental disorders, 5th Edition (DSM-5) (56) as assessed by the Insomnia Interview Schedule
* In the judgment of the investigators and/or consenting professional, able to read and comprehend English
* In the judgment of the consenting professional cognitively able to provide informed consent

Exclusion Criteria:

* As per self report, participant has another sleep disorder provided that it is not adequately treated (e.g., sleep apnea without CPAP treatment)
* As per self report, participant has major depressive disorder, alcohol or drug dependence and
* As per self report, heavy drinker (regularly having more than 14 alcoholic beverages per week)
* As per self report, engaging in night shift work
* To not obscure cortisol assessment, regular smokers per self report (daily use) will be excluded.
* As per self report significant needle phobia as to prevent participation in acupuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
number of participants who complete the assessments | 1 year
  treatment tolerability (rate of CBT-I and acupuncture completion, defined as completing at least 4 out of 7 sessions of CBT-I and 8 out of 10 sessions of acupuncture)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Hunter College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm